CLINICAL TRIAL: NCT04037696
Title: Using a General Health Promotion Approach to Help Smokers With Chronic Diseases Quit: A Randomised Controlled Trial
Brief Title: Using a General Health Promotion Approach to Help Smokers With Chronic Diseases Quit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NTWCREC19001-Main
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive individual face-to-face brief MI (about 5 minutes) on a health-related lifestyle practice. The experimental group will then receive a brief MI via WhatsApp/WeChat on a smartphone during the study period. The brief MI messages will be delivered more intensively as preferred by the subject (usually not less than once every 2 to 3 days and no more than 2 times per day) for the first 6 months. The frequency of delivering the messages via WhatsApp/WeChat will be interactive, depending on the subjects' actions and responses, and may take several sessions of chats within several days or weeks. After 6 months, minimal messages will be provided to the subjects by merely following their progress of behavioural changes and responding to their questions to maintain contact until the 1-year follow-up.
  Interventions: Behavioral: General Health Promotion Approach
- Control group (Other): The control group will be given general brief advice and receive a self-help booklet on smoking cessation published by the Hong Kong Council on Smoking and Health with Hotline will be also provided in the SOPCs. The subjects in this group will receive the same schedule of follow-ups as in the intervention group, but they will not receive any follow-up booster intervention.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: General Health Promotion Approach — The trained Research assistants will ask the subjects about the priority of engaging in any desirable health-related lifestyle practice as identified in the completed baseline questionnaires and to state a targeted goal that they perceive as the easiest to achieve. Each subject will then receive an individual face-to-face brief MI (about 5 mins) with generic health advice on selected health-related lifestyle practice. They will then be informed to receive an individual brief MI intervention to assist behavioural changes or achieve goals as desired or chosen by them via WeChat or WhatsApp in smart phones throughout the study period.
  The RA will then deliver brief MI to each subject individually via WeChat or WhatsApp in smart phones throughout the study period.
  Readiness of quitting smoking will be assessed at 3-month follow-up. Upon request by subjects, we shall provide them with more comprehensive information on quitting.
  Arms: Experimental group
Behavioral: Control — The subjects will be given general brief advice and a self-help smoking cessation booklet with Hotline (Tel.: 1833183). However, subjects in the control group will not receive brief MI and follow-up booster intervention.
  Arms: Control group

SUMMARY:
This study aims to evaluate the effectiveness of a general health promotion (GHP) approach to motivate smokers with chronic diseases to quit smoking. Subjects in the intervention group will receive a brief Motivational Interviewing (MI) using a GHP approach. Subjects in the control group will receive a self-help booklet on smoking cessation at the time of recruitment.

DETAILED DESCRIPTION:
Smoking has harmful effects on nearly every organ of the body and causes seven million deaths worldwide every year. Although the prevalence of daily cigarette smoking in Hong Kong has decreased from 23.3% in 1982 to 10.5 % in 2015, there are still 641,300 daily smokers and 400,000 hospitalisations per year that are attributable to smoking. Having a disease and requiring medical attention present an excellent 'teachable moment' and opportunity for initiating smoking cessation in patients, because they will be more likely to be motivated to alter their habits and improve their health. However, cigarette smoking is addictive and quitting is very difficult, with a high rate of relapse, particularly among patients with chronic diseases.

During the past decade, the investigators have conducted several trials on promoting smoking cessation to smokers with chronic diseases, including cardiac, type 2 diabetes mellitus, and cancer. It is found that many smokers with chronic diseases had a long smoking history, high nicotine dependency, no quit attempt, and no intention to quit. Results of these studies indicated that about 68% smokers with cardiac diseases, 70% with diabetes mellitus and 73% with cancer recruited in Special Out-Patient Clinics (SOPC) were still in the pre-contemplation stage. This revealed that most Hong Kong smokers with chronic diseases perceived more barriers in quitting than the benefits of quitting. Nevertheless, our previous smoking cessation interventions mostly focused on using brief interventions including stage-matched smoking cessation advice. Such interventions could be too brief and inadequate to make a great impact on such smokers. Moreover, the investigators found that using strong warnings to communicate the risk of continued smoking might not be accepted by some of them. Hence, the investigators need to develop and evaluate a more innovative intervention to enhance the effectiveness in promoting smoking cessation for smokers with chronic diseases. Most importantly, the new strategy should have a good potential implementation in many clinical settings.

Smoking has been found to be associated with physical inactivity, unhealthy diet, and drinking. The interrelationship of health behaviours suggests that there could be a higher level of attribute that determines such behaviours together. Our previous studies showed that people with a general intention to promote their health are more likely to engage in desirable health-related lifestyle practices. In addition, research results showed that people once engaged in any desirable health-related lifestyle practices would progressively move to later stages of change for other health behaviours. Based on this concept, a general health promotion approach will be used to motivate smokers with intention to promote health to first engage in any desirable health-related lifestyle practices that are chosen by individual smokers, such as regular physical activity and healthy diet. It is anticipated that once they are engaged in any desirable health-related lifestyle practice they will eventually be more motivated to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above,
* able to speak Cantonese and read Chinese
* no intention to quit smoking (pre-contemplation stage), but are willing to take action to promote health
* have a smart phone and able to use instant messaging tool (e.g. WhatsApp, WeChat) for communication, and
* willing to receive health promotion advices via WhatsApp/WeChat in the smart phone throughout the study

Exclusion Criteria:

* unable to give informed consent or participate in our intervention due to impaired mental status, cognitive impairment, or communication barrier, and
* participation in other smoking cessation programmes or services

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-12-26 (Estimated); Study Completion 2020-12-26 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence at 6 months | 6-month follow-up
  The biochemically validated smoking abstinence will be confirmed by a saliva cotinine level of less than 115 ng/ml in parallel test and a carbon monoxide level in expired air of less than 9 parts per million (ppm)

SECONDARY OUTCOMES:
biochemically validated smoking abstinence at 12 months | 12-month follow-up
  The biochemically validated smoking abstinence will be confirmed by a saliva cotinine level of less than 115 ng/ml in parallel test and a carbon monoxide level in expired air of less than 9 parts per million (ppm)
Self-reported 7-day point prevalence of smoking abstinence at 6 and 12 months | 6- and 12-month follow-up
  A structured questionnaire will be developed by adopting or modifying international and/or locally validated instruments.
Behavioural change | 3-, 6- and 12-month follow-ups
  A structured questionnaire will be developed by adopting or modifying international and/or locally validated instruments.
Smoking quit attempt change from baseline | 3-, 6- and 12-month follow-ups
  A structured questionnaire will be developed by adopting or modifying international and/or locally validated instruments.
Smoking reduction rate change from baseline | 3-, 6- and 12-month follow-ups
  A structured questionnaire will be developed by adopting or modifying international and/or locally validated instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No